CLINICAL TRIAL: NCT03243968
Title: Evaluation of Endothelial and Microvascular Functions in Patients With Myocardial Ischemia Detected by Scintilography and Normal Coronariography
Brief Title: Endothelial and Microvascular Functions in Patients With Myocardial Ischemia
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Camillo L.C. Junqueira (Unknown); Esmeralci Ferreira (Unknown); Maria das Graças C. Souza (Unknown); Eliete Bouskela (Unknown)
Responsible Party: Principal Investigator, Daniel Alexandre Bottino, MD and PHD, Rio de Janeiro State University
Other Study IDs: Biovasc isquêmicos
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Microcirculation; Biomarkers; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic patient - IP: 25 participants with myocardial ischemia detected by scintigraphy and normal coronarography
- Control group - CG: 25 healthy non-ischemic individuals

SUMMARY:
Cardiovascular diseases (CVD) are responsible, throughout the world, for high mortality rates and cardiovascular morbidity. Endothelial dysfunction is the earliest marker of clinical atherosclerosis development. Human studies show that endothelial and microvascular dysfunction are independent predictors of ischemic cardiovascular events and long-term prognosis. The study´s objective is to evaluate the endothelial and peripheral microcirculation changes by venous occlusion plethysmography (VOP), nailfoldvideocapillaroscopy (NVC) and serum biomarkers in patients with myocardial ischemia detected by scintigraphy and normal coronarography.

DETAILED DESCRIPTION:
A cross-sectional study was carried out with 50 participants: 25 with myocardial ischemia detected by scintigraphy and normal coronarography (Ischemic Patient - IP) and 25 healthy non-ischemic individuals (Control Group - CG). All of them were submitted to anamnesis, serum markers (Intercellular Cell Adhesion Molecule [ICAM], Vascular Cell Adhesion Molecule[VCAM], adiponectin, endothelin, LDL-oxidized and CRP-US), NVC and VOP. Exclusion criteria were: inflammatory diseases, cancer patients, recent traumas, Diabetes Mellitus, obese individuals with BMI> 35 kg/m², uncontrolled hypertensive patients, and those with active infectious processes. In the NVC,capillary diameters were observed, as well as red blood cells velocity in the capillaries (RBCV, mm/s), maximum red blood cells after 1 minute ischemia (RBCVmax, mm/s) and time to reach maximal velocity (TRBCVmax) and, regarding VOP,the baseline blood flow (ml/min), post 5 minute ischemia flow and vascular resistance (mmHg/ml/min) were evaluated. Data were analyzed using Student's t-tests for independent or Mann-Whitney samples; χ2 or Fisher exact. The absolute and relative variations (delta) of plethysmography measurements versus baseline in each group were analyzed by the Wilcoxon signed-ranks test and compared between the groups by the Mann-Whitney test. For correction of confounding factors, age and BMI, it was used Covariance Analysis (ANCOVA).

ELIGIBILITY:
Inclusion Criteria:

The study population consisted of 50 patients of both sexes, stratified into two groups: patients with myocardial ischemia detected by scintigraphy (group IP, n = 25) and healthy individuals (CG group, n = 25). In the patients who underwent scintigraphy with tomographic sections and presented any type of image attenuation during the examination, they also underwent a complementary prone position technique. Patients without these characteristics scintigraphy methodologies were excluded from the study.

Exclusion Criteria:

Exclusion criteria were adopted: patients with type 1 or 2 Diabetes Mellitus, heart failure, myocardial infarction or brain stroke with less than three months of the event, chronic renal disease, users of hormonal or non-hormonal anti-inflammatory drugs, recent trauma (less than three months) autoimmune diseases, active infectious processes, presence of neoplasia, use of Aspirin (anti-inflammatory dose), obesity with BMI>35 kg/m², uncontrolled hypertensive patients, resistant hypertensives, and non-compliance in the examinations or with the signature of the Consent Form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty patients were studied: 39% male and 61% female. The mean age was 48 ± 15.8 years, being: 56.5 ± 10.5 years in the IP group and 39.4 ± 15.8 years in the CG. The mean BMI was 26.5 ± 4.30 kg/m².
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
%Hyper | One year
  Increment of forearm blood flow during reactive hyperemia after 5 minutes arm ischemia with venous occlusion plethysmography.

SECONDARY OUTCOMES:
Intercellular adhesion molecule (ICAM) | One year
  Inflammatory biomarker obtained through withdrawal of venous blood.
Vascular adhesion molecule (VCAM) | One year
  Inflammatory biomarker obtained through withdrawal of venous blood.
Adiponectin | One year
  Adipokyne obtained through withdrawal of venous blood.
Endothelin | One year
  Potent vasoconstrictor obtained through withdrawal of venous blood.
LDL-oxidized | One year
  Low density lipoprotein oxidized used to measure oxidative stress. It is obtained from venous blood.
CRP | One year
  C reactive protein obtained through withdrawal of venous blood.
% Nitro | One year
  Increment of forearm blood flow after 5 minutes of 400 μg sublingual nitroglycerin application with venous occlusion plethysmography..
FCD | One year
  Functional capillary density. Number of capillaries with flowing red blood cell in microscope area. Obtained from Nailfold videocapillaroscopy.
AFCD | One year
  Afferent capillar diameter. Obtained from Nailfold videocapillaroscopy.
ACD | One year
  Apical capillar diameter. Obtained from Nailfold videocapillaroscopy.
EFCD | One year
  Efferent capillar diameter. Obtained from Nailfold videocapillaroscopy.
RBCV | One year
  Basal red blood cell velocity. Obtained from Nailfold videocapillaroscopy.
RBCVmax | One year
  Maximum red blood cell velocity during reactive hyperemia in fourth finger after one minute ischemia. Obtained from Nailfold videocapillaroscopy.
TRBCVmax | One year
  Time to reach Maximum red blood cell velocity during reactive hyperemia in fourth finger after one minute ischemia. Obtained from Nailfold videocapillaroscopy.
%ResHyper | One year
  Increment of vascular resistance during reactive hyperemia after 5 minutes arm ischemia with venous occlusion plethysmography.
%ResNitro | One year
  Increment of vascular resistance after 5 minutes of 400 μg sublingual nitroglycerin application with venous occlusion plethysmography.

IPD SHARING:
Plan to Share IPD: No